CLINICAL TRIAL: NCT06238908
Title: Clinical Study on the Safety and Efficacy of an Intravenous Infusion of NGGT003 in the Treatment of Hemophilia A
Brief Title: Safety and Efficacy Study of NGGT003 in Hemophilia A Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023043
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 3 doses of NGGT003 will be administered according to the principle of dose escalation
  Interventions: Drug: NGGT003

INTERVENTIONS:
Drug: NGGT003 — Single intravenous infusion of NGGT003 at low dose (4e11vg/kg), medium dose (1e12vg/kg) and high dose (2.5e12vg/kg)

SUMMARY:
This is an early phase 1, open-label, single-center, dose-escalation pilot trial to evaluate the safety and efficacy of an intravenous infusion of NGGT003 in hemophilia A patients. NGGT003 uses adeno-associated virus (AAV) as a vector, carrying a liver specific promoter and codon optimized human FVIII gene B domain deletion mutant (hFVIII BDD), and expresses human FVIII protein in the liver through intravenous injection.

DETAILED DESCRIPTION:
Hemophilia A (HA) is an X-linked recessive genetic disease caused by mutations in the FVIII gene on the X chromosome, leading to abnormal coagulation function. In the male population, the incidence rate of hemophilia A was about 1/5000, and female patients with hemophilia A were extremely rare. Type A hemophilia patients mainly exhibit a tendency for bleeding, with a wide range of bleeding sites and frequent recurrence, which can form hematoma and joint deformation. This is an early phase 1, open-label, single-center, dose-escalation pilot trial to evaluate the safety and efficacy of a single intravenous infusion of NGGT003 in hemophilia A patients. 4-6 subjects will be enrolled and divided into 3 groups according to the principle of dose escalation, respectively administered intravenous infusion of NGGT003 at low dose (4e11vg/kg), medium dose (1e12vg/kg) and high dose (2.5e12vg/kg). All subjects will undergo 52 weeks of treatment observation and further 260 weeks of long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. Male, age ≥18 years old;
3. Diagnosed with hemophilia A according to the "Guidelines for Diagnosis and Treatment of Hemophilia A (2022 Edition)", and the endogenous FVIII activity level was <1 IU/dL (<1%);
4. The exposure days (EDs) of treatment with any recombinant or plasma-derived FVIII product were ≥150 days;
5. Anti-AAV neutralizing antibody titer ≤1:5, binding antibody titer ≤1:100;
6. Bleeding events and/or FVIII product injections have occurred within 12 weeks before screening;
7. No history of allergy to FVIII products;
8. FVIII inhibitor titer﹤0.6BU/mL;
9. Commitment to use other drugs during the study requires the consent of the investigator;
10. Willing and able to comply with study procedures and requirements;
11. Willing to use effective contraceptive methods within 52 weeks after administration.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen, hepatitis C, human immunodeficiency virus (HIV)，syphilis test;
2. Clinically significant abnormalities in liver function test: alanine aminotransferase (ALT) >1.5 × upper limit of normal (ULN) and/or aspartate aminotransferase (AST) >1.5× ULN;TBil）>1.5×ULN；Serum creatinine (Scr) >1.5×ULN; hemoglobin <110g/L, platelets <10e9/L;
3. History of being positive for FVIII inhibitors;
4. Have other bleeding factors except hemophilia;
5. Plan major surgery within 52 weeks;
6. Have contraindications to glucocorticoid, including but not limited to allergy to glucocorticoids, epilepsy, new unhealed fractures, in trauma repair period, uncontrolled infection, severe osteoporosis, etc, which assessed and determined by the investigators;
7. History of allergy to human albumin;
8. Have serious diseases or active infections in cardiovascular, respiratory, digestive tract, endocrine, renal, blood, nervous, mental and other systems before screening;
9. With hepatitis, cirrhosis, liver cancer or other major liver diseases;
10. History of malignant tumors;
11. Abnormal and clinical significant vital signs, physical examination, laboratory examination or other related examination results during the screen, which are not suitable for trial according to the investigator;
12. Previous gene therapy treatment;
13. Participation in any other clinical trial before the screening and have taken medication within four weeks or five half-lives of the study drug;
14. Any other condition that may not be appropriate for the study in the opinion of the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) | 52 weeks
  Incidence of AE and SAE, as assessed by physical examinations, clinical laboratory parameters and adverse event reporting
Changes in annualized bleeding rate (ABR) | 52 weeks
  Changes in annualized bleeding rate (ABR) from baseline to 52 weeks.

SECONDARY OUTCOMES:
FVIII activity levels | 52 weeks
  Change in FVIII activity levels from baseline to week 52.
FVIII protein product infusions | 52 weeks
  Calculate the number and volume of FVIII protein product infusions from baseline to week 52.
Target joints | 52 weeks
  Changes the numbers of target joints from baseline to week 52.
HA-QOL scores | 52 weeks
  Change in HA-QOL scores from baseline to 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No